CLINICAL TRIAL: NCT01935830
Title: Efavirenz and Ritonavir Influence on Human Brain Levo-acetylmethadol (LAAM) Disposition Assessed Using PET Imaging
Brief Title: LAAM-HAART PET Imaging
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201307040
Record Dates: First submitted 2013-08-30; First posted 2013-09-05 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Healthy Volunteers
Keywords: PET Imaging; Efavirenz; Ritonavior [11C] LAAM; Healthy volunteers
MeSH Terms: interventions — Methadyl Acetate; Ritonavir; lopinavir-ritonavir drug combination; efavirenz; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LAAM arm (Experimental): 1. [11C]LAAM 15-20 mCi (maximum administered mass of 10 ug)
  2. Efavirenz, oral capsules, 600 mg
  3. Ritonavir, oral capsules, 100 mg
  Interventions: Radiation: [11c] LAAM; Drug: Ritonavir; Drug: Efavirenz

INTERVENTIONS:
Radiation: [11c] LAAM — intravenous administration of 15-20 mCi of [11c] LAAM.
Drug: Ritonavir — Pretreatment with oral ritonavir for 3 days followed by intravenous administration of 15-20 mCI of [11c] LAAM.
  Other Names: Kaletra
Drug: Efavirenz — Pretreatment with oral Efavirenz 600 mg orally every night x 14 days followed by intravenous administration of 15-20 mCI of [11c] LAAM.
  Other Names: Sustiva, Atripla

SUMMARY:
The purpose of this study is to determine the effects of the antiretroviral drugs efavirenz and ritonavir on human brain LAAM disposition in vivo.

ELIGIBILITY:
Inclusion

Each subject must meet all of the following criteria:

1. Male or non-pregnant female volunteer, 18-50 yr old
2. Good general health with no known major medical conditions
3. BMI < 33
4. Provide informed consent

Exclusion Criteria

Subjects will not be enrolled if any of the following criteria exist:

1. Known history of liver or kidney disease
2. History of major medical conditions
3. HIV seropositive
4. Fasting blood glucose > 110 mg/dl (because HAART can cause glucose intolerance)
5. Family history of type 2 diabetes
6. Use of prescription or non prescription medications, herbals or foods known to be metabolized by or altering P-glycoprotein or CYP3A (hormonal birth control medications are acceptable if alternative means of contraception are used)
7. Females who are pregnant or nursing
8. Females taking hormonal contraceptives who are unwilling to use alternative means of contraception
9. Contraindications to MRI (e.g., metal implants or splinters in the body; a worn or implanted medical device, such as a pacemaker or drug pump; inability to lie flat for up to one hour; claustrophobia) or contraindications to PET scanning (e.g., inability to lie flat for up to one hour, claustrophobia, current
10. Current or recent (within 12 months prior to screening) participation in research studies involving radiation exposure such that the total research-related radiation dose to the subject in any given year would exceed the limits set forth in the US Code of Federal Regulations (CFR) Title 21 Section 361.1 (http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/CFRSearch.cfm?FR=361.1))

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
cerebral [11C]LAAM distribution volume | approximately 3 months
  Blood tests, MRI and PET data analysis and interpretation

CONTACTS AND LOCATIONS:
Overall Officials: Evan D Kharasch, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No